CLINICAL TRIAL: NCT03241199
Title: A Phase II Study to Determine the Efficacy and Safety of Induction-Maintenance Protocol for Patients With Chronic-Phase Chronic Myelogenous Leukaemia
Brief Title: The Efficacy and Safety of Induction-Maintenance Protocol for Patients With Chronic Myelogenous Leukaemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Yok-lam Kwong, Chair Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QMH-CML-002
Record Dates: First submitted 2017-08-02; First posted 2017-08-07 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Chronic Myeloid Leukemia; Philadelphia Chromosome Positive CML
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imatinib Mesylate (Experimental): imatinib 400mg daily
  Interventions: Drug: Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib Mesylate — a first-generation tyrosine kinase inhibitors

SUMMARY:
The purpose of this pilot study is to investigate whether some patients who were started on a 2G-TKI as first-line treatment can be safely switched to imatinib, a first-generation TKI, while maintaining or even deepening the molecular response as a cost-effective treatment. Eligible patients will be switched to imatinib 400mg daily, with regular molecular monitoring.

DETAILED DESCRIPTION:
Imatinib, nilotinib and dasatinib are standard first-line options for newly diagnosed patients with chronic-phase chronic myeloid leukemia (CML). While nilotinib and dasatinib, also known as second-generation TKI (2G-TKI), have been shown to result in earlier and deeper molecular response, they have not been proven superior to imatinib in terms of clinical outcomes like progression-free survival and overall survival. Moreover, their long-term safety has been questioned: nilotinib is associated with increased cardiovascular risk while dasatinib causes pleural effusion in significant proportion of patients and may even lead to pulmonary hypertension.

The purpose of this pilot study is to investigate whether some patients who were started on a 2G-TKI as first-line treatment can be safely switched to imatinib, a first-generation TKI, while maintaining or even deepening the molecular response as a cost-effective treatment. Eligible patients will be switched to imatinib 400mg daily, with regular molecular monitoring.

In case of molecular progression

The following should be systematically performed:

* Clinical examination
* Baseline blood test including complete blood count (CBC), liver and renal function, lactate dehydrogenase (LDH), urate
* Restart the original 2G-TKI and in same dose as given before study entry unless medically indicated to change therapy
* Screening of breakpoint cluster region- Abelson murine leukemia (BCR-ABL) kinase domain mutations
* In the absence of signs of haematological relapse or breakpoint cluster region- Abelson murine leukemia (BCR-ABL1) ≥ 1% (IS ratio), bone marrow aspiration and cytogenetics are not routinely performed unless deemed indicated by the physician in charge.

The patient will be followed until major molecular response (MMR) is re-achieved and further 6 months beyond. Date of progression, hematological data at progression (molecular, cytogenetic, and hematological), and treatment proposed for molecular progression and response to it (molecular, cytogenetic, hematological) will be collected. Follow-up for overall survival (OS) and progression-free survival (PFS) will last 2 years since the date of switch of TKI.

In case of loss of complete hematological response (CHR) or any sign of accelerated or blastic phase of CML, the patient will be immediately considered as in disease progression and TKI should be started immediately.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (aged 18 years or above) patients diagnosed with chronic-phase CML
2. Must have received a 2G-TKI (nilotinib or dasatinib) as first-line therapy for at least 12 months (Note: Cytoreductive agents, namely hydroxyurea and anagrelide, prior to the use of TKI are allowed.)
3. In sustained, good molecular response (i.e. molecular response (MR3) or below) for at least 6 months, as confirmed with at least 2 consecutive quantitative real time-polymerase chain reaction (RT-PCR) results

Exclusion Criteria:

1. Under 18 years old
2. Adults under law protection or without ability to consent
3. Previous or planned autologous/allogeneic haematopoietic stem cell transplantation
4. Documented kinase domain mutation
5. A change to the current TKI because of unsatisfactory response to a previous TKI (Note: patients are still considered eligible if the switch in TKI was due to intolerance or side effects)
6. History of disease progression (accelerated or blast phase)
7. Patients who can speak neither Chinese nor English
8. Any molecular result during the preceding 6 months that is higher than MR3, i.e. BCR-ABL1/ABL1 ratio >0.1% on IS ratio

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-06-13 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
molecular progression-free survival | 6 months
  Molecular progression-free survival after switch to imatinib at 6 months

SECONDARY OUTCOMES:
molecular progression-free survival | 12 months
  Molecular progression-free survival after switch to imatinib at 12 months
molecular progression-free survival | 24 months
  Molecular progression-free survival after switch to imatinib at 24 months
Molecular responses | 12 months
  Molecular responses after switch to imatinib at 12 months
Molecular responses | 24 months
  Molecular responses after switch to imatinib at 24 months
Rate of molecular progression on Imatinib | 24 months
  Number of patients who have molecular progression on Imatinib
Rate of regain MMR after resumption of original TKI and time to recovery of MMR | 24 months
  Number of patients who regain MMR on resumption of their original TKI, and time to recovery of MMR

CONTACTS AND LOCATIONS:
Overall Officials: Carol Cheung, MBBS, Principal Investigator — Queen Mary Hospital, Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided